CLINICAL TRIAL: NCT03718039
Title: A Phase 2 Open-Label Study of HTX-011 Via Individualized Dosing Administration for Postoperative Analgesia Following Unilateral Simple Bunionectomy
Brief Title: Phase 2 Bunionectomy HTX-011 Administration Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HTX-011-218
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Pain
Keywords: bunion; bunionectomy; bunion surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Bunion | interventions — Aprepitant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Treatment Group 1: HTX-011 (Experimental): HTX-011 (bupivacaine/meloxicam), up to but not to exceed 60 mg/1.8 mg, via instillation.
  Interventions: Drug: HTX-011; Device: Luer Lock applicator; Device: Vial access device
- Treatment Group 2: HTX-011 + Aprepitant (Experimental): HTX-011 (bupivacaine/meloxicam), up to but not to exceed 60 mg/1.8 mg, via instillation; Aprepitant, three single doses of aprepitant will be administered orally.
  Interventions: Drug: HTX-011; Device: Luer Lock applicator; Device: Vial access device; Drug: aprepitant
- Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen (Experimental): HTX-011 (bupivacaine/meloxicam), up to but not to exceed 60 mg/1.8 mg, via instillation and a scheduled multimodal analgesic (MMA) regimen.
  Interventions: Drug: HTX-011; Device: Luer Lock applicator; Device: Vial access device

INTERVENTIONS:
Drug: HTX-011 — HTX-011 (bupivacaine/meloxicam), up to but not to exceed 60 mg/1.8 mg, via instillation.
Device: Luer Lock applicator — Applicator for instillation.
Device: Vial access device — Device for withdrawal of drug product.
Drug: aprepitant — Aprepitant, three single doses of aprepitant will be administered orally.
  Arms: Treatment Group 2: HTX-011 + Aprepitant

SUMMARY:
This is a Phase 2, open-label, multi-cohort study to evaluate the analgesic efficacy, safety, and pharmacokinetics (PK) of a single, individualized dose of HTX-011 administered into the surgical site as a monotherapy or with other medications to enhance analgesia in subjects undergoing unilateral simple bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo a primary unilateral, distal, first metatarsal bunionectomy with osteotomy and internal fixation under regional anesthesia.
* Has an American Society of Anesthesiologists Physical Status of I, II, or III.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or using acceptable contraceptives. For cohort 2, acceptable contraceptives excludes hormonal contraceptives.

Exclusion Criteria:

* Has had a contralateral foot bunionectomy in the past 3 months prior to the scheduled surgery.
* Has a planned concurrent surgical procedure (eg, bilateral bunionectomy or collateral procedures on the surgical foot).
* Has a pre-existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
* Has taken any NSAIDs within at least 10 days prior to the scheduled surgery.
* Has taken long-acting opioids within 3 days prior to the scheduled surgery.
* Has taken any opioids within 24 hours prior to the scheduled surgery.
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* For Cohort 2 only, has been administered aprepitant or another NK1 receptor antagonist within 5 days prior to the scheduled surgery.
* Has been administered any local anesthetic within 72 hours prior to the scheduled surgery.
* Has initiated treatment with study medications within 1 month prior to study drug administration that can impact pain control.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of study drug.
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* As per subject history and/or medical records, has active infection or is currently undergoing treatment for Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV).
* Has uncontrolled anxiety, psychiatric, or neurological disorder.
* For Cohort 2 only, is receiving pimozide, a strong or moderate CYP3A4 inhibitor, or a strong CYP3A4 inducer.
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse. Note: Subjects with a positive drug screen who are taking an allowed, prescribed medication that is known to result in a positive drug test (eg, amphetamine and dextroamphetamine for attention-deficit/hyperactivity disorder, benzodiazepine for anxiety disorder) may be eligible for participation in the study at the discretion of the Sponsor. Subjects taking any marijuana (medical or recreational) are not allowed to participate in the study.
* Previously participated in an HTX-011 study.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half-lives.
* Has undergone 3 or more surgeries within 12 months.
* Has a body mass index (BMI) >39 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Endeavor Clinical Trials, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: HTX-011 + Aprepitant | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen
Started | 30 | 17 | 31
Completed | 30 | 17 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: HTX-011 + Aprepitant | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen | Total
Number analyzed (Participants) | 30 | 17 | 31 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 16 | 29 | 75
  >=65 years | 0 | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (11.58) | 43.7 (14.73) | 49.1 (12.66) | 47.2 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 13 | 29 | 70
  Male | 2 | 4 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 12 | 15 | 42
  Not Hispanic or Latino | 15 | 5 | 16 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 4 | 6
  White | 28 | 16 | 27 | 71
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 17 | 31 | 78

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve (AUC) of the NRS-A (Windowed Worst Observation Carried Forward) Pain Intensity Scores
Description: Pain intensity scores are assessed using an 11-point Numeric Rating Scale (NRS) (0-10) where 0 represents "no pain" and 10 represents "worst pain imaginable". NRS scores are recorded with activity (NRS-A), sitting with the plantar surface of the ball of the surgically attended foot touching the floor (no weight-bearing).
Time Frame: 72 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: HTX-011 + Aprepitant | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen
Number analyzed (Participants) | 30 | 17 | 31
pain intensity score*hr | 278.36 (151.085) | 288.23 (115.790) | 126.93 (129.819)

2. Secondary Outcome: Mean Total Postoperative Opioid Consumption (in Morphine Equivalents) Through 72 Hours
Time Frame: 72 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: MME, morphine milligram equivalents
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: HTX-011 + Aprepitant | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen
Number analyzed (Participants) | 30 | 17 | 31
MME, morphine milligram equivalents | 11.47 (10.198) | 21.88 (13.305) | 1.61 (3.449)

3. Secondary Outcome: Percentage of Subjects Receiving no Opioid Rescue
Time Frame: 72 hours
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: HTX-011 + Aprepitant | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen
Number analyzed (Participants) | 30 | 17 | 31
Participants | 6 | 0 | 24

4. Secondary Outcome: Percentage of Subjects Receiving no Opioid Rescue
Description: Only subjects in Cohort 3 received a scheduled, non-opioid MMA regimen following surgery.
Time Frame: Day 7 and Day 28
Population: Safety Population, Cohort 3 only
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen
Number analyzed (Participants) | 31
Participants
  Day 7 | 24
  Day 28 | 24

5. Secondary Outcome: Mean Area Under the Curve (AUC) of the NRS-R (Windowed Worst Observation Carried Forward) Pain Intensity Scores
Description: Pain intensity scores are assessed using an 11-point Numeric Rating Scale (NRS) (0-10) where 0 represents "no pain" and 10 represents "worst pain imaginable". NRS scores are measured at rest.
Time Frame: 72 hours
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: HTX-011 + Aprepitant | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen
Number analyzed (Participants) | 30 | 17 | 31
pain intensity score*hr | 251.92 (127.319) | 252.39 (112.996) | 113.10 (124.696)

ADVERSE EVENTS:
Time Frame: 42 Days.
Description: For each PT, subjects are included only once, even if they experienced multiple events in that PT.
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: HTX-011 + Aprepitant | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/17 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/17 | 0/31
Other Adverse Events (participants affected / at risk) | 13/30 | 13/17 | 16/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1: HTX-011 (N=30) | Treatment Group 2: HTX-011 + Aprepitant (N=17) | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen (N=31)
Cellulitis (Infections and infestations) | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1: HTX-011 (N=30) | Treatment Group 2: HTX-011 + Aprepitant (N=17) | Treatment Group 3: HTX-011 + Non-Opioid MMA Regimen (N=31)
Localised infection (Infections and infestations) | 0 | 0 | 2
Tinea pedis (Infections and infestations) | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 6 | 7
Constipation (Gastrointestinal disorders) | 0 | 5 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT03718039/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT03718039/SAP_001.pdf